CLINICAL TRIAL: NCT03318939
Title: A Phase 2 Study of Poziotinib in Patients With Non-Small Cell Lung Cancer (NSCLC), Locally Advanced or Metastatic, With EGFR or HER2 Exon 20 Insertion Mutation (ZENITH20)
Brief Title: Phase 2 Study of Poziotinib in Participants With NSCLC Having EGFR or HER2 Exon 20 Insertion Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision (unrelated to safety)
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-202
Record Dates: First submitted 2017-10-10; First posted 2017-10-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: NSCLC
Keywords: EGFR; HER2; Exon 20 insertion mutation
MeSH Terms: interventions — HM781-36B

STUDY DESIGN:
Intervention Model Description: Each treatment cycle is 28 calendar days in duration. There will be seven participant cohorts and eligible participants will be enrolled into each cohort in parallel based on EGFR or HER2 exon 20 mutation status and prior treatment status:
  * Cohort 1: Previously treated participants with EGFR exon 20 insertion mutant positive NSCLC (closed to enrollment)
  * Cohort 2: Previously treated participants with HER2 exon 20 insertion mutant positive NSCLC (closed to enrollment)
  * Cohort 3: Treatment naïve participants with EGFR exon 20 insertion mutant positive NSCLC (fully enrolled)
  * Cohort 4: Treatment naïve participants with HER2 exon 20 insertion mutant positive NSCLC
  * Cohort 5: Participants who meet the criteria for enrollment in Cohort 1 to 4, but the enrollment in the respective cohort has been closed
  * Cohort 6: Participants with acquired EGFR mutation who progressed while on treatment with first-line osimertinib
  * Cohort 7: Participants with EGFR or HER2 activating mutations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poziotinib (Experimental): * Cohort 1: Previously treated participants with EGFR exon 20 insertion mutant positive NSCLC (closed to enrollment)
  * Cohort 2: Previously treated participants with HER2 exon 20 insertion mutant positive NSCLC (closed to enrollment)
  * Cohort 3: Treatment naïve participants with EGFR exon 20 insertion-mutant positive NSCLC (fully enrolled)
  * Cohort 4: Treatment naïve participants with HER2 exon 20 insertion mutant positive NSCLC
  * Cohort 5: Participants who meet the criteria for enrollment in Cohort 1 to 4, but the enrollment in the respective cohort has been closed
  * Cohort 6: Participants with acquired EGFR mutation who progressed while on treatment with first-line osimertinib
  * Cohort 7: Participants with EGFR or HER2 activating mutations
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — The poziotinib drug substance is a hydrochloride salt of poziotinib and is formulated as a tablet for oral administration.
  * Cohorts 1-3: 16 mg QD
  * Cohort 4: 8 mg BID
  * Cohort 5: randomized to 8 mg BID or 6 mg BID or 10 mg QD
  * Cohorts 6 and 7: 8 mg BID

SUMMARY:
This is a Phase 2, open-label, multi-center study to evaluate the efficacy and the safety/tolerability of poziotinib in seven participant cohorts for up to 603 previously treated and treatment-naïve NSCLC participant. Cohorts 3 and 4 were added with Amendment 1 and three additional cohorts were added with Amendment 2 (Cohorts 5, 6 and 7).

DETAILED DESCRIPTION:
The Screening period (Day -30 to Day -1) lasts up to approximately 30 days prior to Cycle 1, Day 1. Participant must meet all Inclusion/Exclusion Criteria to participate in the study. Eligible participants will provide written Informed Consent prior to undergoing any study procedures.

Each treatment cycle is 28 calendar days in duration. There will be seven participant cohorts and eligible participants will be enrolled into each cohort in parallel based on EGFR or HER2 exon 20 mutation status and prior treatment status:

* Cohort 1: Previously treated participant with EGFR exon 20 insertion mutation positive NSCLC (complete)
* Cohort 2: Previously treated participant with HER2 exon 20 insertion mutation positive NSCLC (complete)
* Cohort 3: Treatment naïve participant with EGFR exon 20 insertion mutation positive NSCLC (complete)
* Cohort 4: Treatment naïve participant with HER2 exon 20 insertion mutation positive NSCLC (fully enrolled)
* Cohort 5: Participants who meet the criteria for enrollment in Cohort 1 to 4, but the enrollment in the respective cohort has been closed (closed to enrollment)
* Cohort 6: Participants with acquired EGFR mutation who progressed while on treatment with first-line osimertinib (closed to enrollment)
* Cohort 7: Participants with EGFR or HER2 activating mutations (closed to enrollment)

Toxicity will be assessed based on the grade of the adverse events using CTCAE version 4.03.

On Day 1 of each 28-day cycle, the participant's absolute neutrophil count (ANC) must be ≥1.5×10^9/L and platelet count must be ≥100×10^9/L before administering poziotinib. All participants will be treated until disease progression (except for first progression in Cohort 5), death, intolerable adverse events (AEs), or other protocol-specified reasons for participant withdrawal.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must be willing and capable of giving written Informed Consent, adhering to dosing and visit schedules, and meeting all study requirements
* Participant has histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) that is not amenable to treatment with curative intent
* Prior treatment status:

  * Cohorts 1 and 2: Participant has had at least one prior systemic treatment for locally advanced or metastatic NSCLC
  * Cohorts 3 and 4: Participant is treatment-naïve for locally advanced or metastatic NSCLC and eligible to receive first-line treatment with poziotinib as determined by the Investigator. Adjuvant/neo-adjuvant therapies (chemotherapy, radiotherapy, or investigational agents) are permissible as long as they end at least 15 days prior to study entry.
  * Cohort 5: Participants who meet the criteria for enrollment in Cohorts 1 to 4, but the enrollment in the respective cohort has been closed
  * Cohort 6: Participant with EGFR mutation-positive NSCLC who progressed while on treatment with first-line osimertinib
  * Cohort 7: Participant has had at least one prior systemic treatment for locally advanced or metastatic NSCLC
* Specific mutations:

  * Cohort 1 and 3: Documented EGFR exon 20 insertion mutation
  * Cohort 2 and 4: Documented HER2 exon 20 insertion mutation
  * Cohort 5: Documented EGFR or HER2 exon 20 insertion mutations
  * Cohort 6: Documented acquired EGFR mutation (tested after osimertinib progression)
  * Cohort 7: Documented EGFR or HER2 activating mutations
* Participant has adequate organ function at Baseline

Key Exclusion Criteria:

* Participant has had previous treatment with poziotinib or any other EGFR or HER2 exon 20 insertion mutation-selective tyrosine kinase inhibitor (TKI) prior to study participation. The currently approved TKIs (ie, erlotinib, gefitinib, afatinib, osimertinib) are not considered to be exon 20 insertion-selective and are permissible (Cohorts 1 and 2).
* Participant is concurrently receiving chemotherapy, biologics, immunotherapy for cancer treatment; systemic anti-cancer treatment or investigational treatment should not be used within 2 weeks or 5 half lives, whichever is longer; local radiation therapy for bone pain may be allowed
* Participant has had other malignancies within the past 3 years, except for stable non-melanoma skin cancer, fully-treated and stable, early-stage prostate cancer, or carcinoma in situ of the cervix or breast without need of treatment
* Participant is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of poziotinib to the end of study.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  The proportion of subjects who achieve CR, PR, and Stable Disease (SD) by the best response from the first dose of poziotinib to the end of study.
Duration of Response (DoR) | 24 months
  Number of days from the date that measurement criteria are first met for CR or PR (whichever status is recorded first) until the first subsequent date that progressive disease or death is documented.

OTHER OUTCOMES:
Progression-free Survival (PFS) - Exploratory | 24 months
  Number of days from the treatment start date to the date of documented disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (63):
- United States (43):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Oncology Physician's Network Inc./OPN Healthcare, Arcadia, California
  - City of Hope, Duarte, California
  - UCSD -Moores Cancer Center, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Helen Diller Comprehensive Cancer Center at Mt Zion, San Francisco, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - Yale University, Yale Cancer Center Smilow Cancer Hospital at Yale, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The Bond & Steele Clinic, P.A. dba Bond Clinic, P.A., Winter Haven, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - CTCA - Southeastern Regional Medical Center, Newnan, Georgia
  - CTCA - Midwestern Regional Medical Center, Zion, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - North Shore Hematology Oncology Associates P.C. DBA NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - Montefiore Einstein Medical Center for Cancer Care, The Bronx, New York
  - North Shore Hematology Oncology Associates DBA New York Cancer and Blood Specialists, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - CTCA - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology- Austin, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (4):
  - Saint Luc University Hospital, Brussels
  - University Hospitals Leuven, Leuven
  - Ambroise Pare University Hospital Center, Mons
  - General Hospital Delta, Roeselare
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (2):
  - Hopital Larrey, CHU Toulouse, Unité d'Oncologie des Voies Respiratoires, Toulouse
  - Gustave Roussy Oncology Institute, Department of Medical Oncology, Villejuif
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Healthcare Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (3):
  - National Cancer Institute, IRCCS, Department of Medical Oncology, Milan
  - Santa Maria delle Croci Hospital, Ravenna
  - National Cancer Institute Regina Elena, IRCCS, Operative Unit of Medical Oncology A 1, Rome
- Erasmus Medical Center, Rotterdam, Netherlands
- Spain (2):
  - University Hospital Germans Trias i Pujol, Department of Medical Oncology, Barcelona
  - University Hospital 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le X, Cornelissen R, Garassino M, Clarke JM, Tchekmedyian N, Goldman JW, Leu SY, Bhat G, Lebel F, Heymach JV, Socinski MA. Poziotinib in Non-Small-Cell Lung Cancer Harboring HER2 Exon 20 Insertion Mutations After Prior Therapies: ZENITH20-2 Trial. J Clin Oncol. 2022 Mar 1;40(7):710-718. doi: 10.1200/JCO.21.01323. Epub 2021 Nov 29. PMID 34843401